CLINICAL TRIAL: NCT03360435
Title: Absorption of Transdermal Vitamins in Post Bariatric Surgery Patients
Status: Completed | Type: Observational
Sponsor: University of Florida (Other)
Responsible Party: Sponsor
Other Study IDs: IRB201701809
Record Dates: First submitted 2017-11-17; First posted 2017-12-04 (Actual); Last update posted 2021-07-09 (Actual); Status verified 2021-07

CONDITIONS: Bariatric Surgery Candidate; Vitamin Deficiency; Mineral Deficiency
MeSH Terms: conditions — Avitaminosis | interventions — Transdermal Patch

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Participants with transdermal patches: All study subjects will belong to the same group. This group will undergo bariatric surgery and will use a transdermal patch for vitamin and mineral supplementation post operatively. The transdermal patch will be the Patch MD MultiVitamin Plus patch
  Interventions: Dietary Supplement: Patch MD MultiVitamin Plus patch

INTERVENTIONS:
Dietary Supplement: Patch MD MultiVitamin Plus patch — The transdermal patch contains vitamins A, D, E, K2, C, thiamine, riboflavin, niacin, pantothenic acid, pyridoxine, biotin, folic acid, cyanocobalamin, calcium, iron, phosphorous, iodine, magnesium, zinc, selenium, copper, manganese, chromium, molybdenum, potassium, chloride, and boron.

SUMMARY:
Patients undergoing bariatric surgery often develop new vitamin and/or mineral deficiencies or exacerbate prior deficiencies after surgery. Several bariatric supplement products exist including oral tablets and transdermal patches. The purpose of this study is to observe the concentrations of serum micronutrients and determine how many deficiencies develop in patients who use a transdermal patch.

DETAILED DESCRIPTION:
Patients will undergo either a sleeve gastrectomy or gastric bypass procedure. All patients enrolled will have previously chosen to use the Patch MD MultiVitamin Plus patch for vitamin and mineral supplementation versus oral or other dosage forms of vitamins after surgery. A conversation between the patient and provider will occur first during a pre operative appointment, at which time the patient will be presented with the option to use oral vitamins or the Patch MD MultiVitamin Plus patch after surgery. Only if the patient chooses the patch will he/she be made aware of the study and recruited. Pre operative blood draws will be used to determine baseline micronutrient serum concentrations and existing deficiencies. The Gastrointestinal Symptom Rating Scale (GSRS) will be used pre operatively to determine baseline gastrointestinal symptoms. Post operative blood draws and GSRS data will be collected at 3 months, 6 months, and 1 year after surgery.

ELIGIBILITY:
Inclusion Criteria:

1. Candidates for a sleeve gastrectomy or gastric bypass surgery
2. Willingness and ability to provide informed consent in English
3. Commitment to the 1 year study period

Exclusion Criteria:

1. Planned bariatric revision surgery
2. Patients with a left ventricular assistance device
3. Known End Stage Renal Disease
4. Known mutation in methylenetetrahydrofolate reductase (MTHFR) gene
5. Medical conditions requiring vitamin and mineral supplementation

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Adult patients undergoing bariatric surgery for weight loss who have chosen to use a transdermal patch for vitamin and mineral supplementation will be recruited to complete the study. All eligible patients within the institution will be recruited.
Sampling Method: Non-Probability Sample
Enrollment: 99 (Actual)
Dates: Start 2017-12-15 (Actual); Primary Completion 2021-07-07 (Actual); Study Completion 2021-07-07 (Actual)

PRIMARY OUTCOMES:
Percentage of subjects with deficiencies | 1 year
  The primary end point is the percentage of participants who have two or more deficiencies of vitamins B1, B6, B12, folate, D, zinc, calcium, copper, and iron one year after bariatric surgery after using the Patch MD™ MultiVitamin Plus transdermal patch for supplementation.

SECONDARY OUTCOMES:
Thiamine | 1 year
  The average decrease in the serum concentration among all subjects
Pyridoxine | 1 year
  The average decrease in the serum concentration among all subjects
Methylcobalamin | 1 year
  The average decrease in the serum concentration among all subjects
Vitamin D | 1 year
  The average decrease in the serum concentration among all subjects
Folate | 1 year
  The average decrease in the serum concentration among all subjects
Zinc | 1 year
  The average decrease in the serum concentration among all subjects
Calcium | 1 year
  The average decrease in the serum concentration among all subjects
Copper | 1 year
  The average decrease in the serum concentration among all subjects
Iron | 1 year
  The average decrease in the serum concentration among all subjects
Ferritin | 1 year
  The average decrease in the serum concentration among all subjects
Parathyroid hormone | 1 year
  The average decrease in the serum concentration among all subjects
Total iron binding capacity | 1 year
  The average decrease among all subjects
Constipation syndrome | 1 year
  The average increase among all subjects using the Gastrointestinal Symptom Rating Scale. For constipation syndrome, three symptoms (constipation, hard stools, feeling of incomplete evacuation) will each be measured on a seven point Likert scale (0=no symptom, 6=most severe symptom). The three values will be averaged to provide one value which will represent constipation syndrome.
Diarrhea syndrome | 1 year
  The average increase among all subjects using the Gastrointestinal Symptom Rating Scale. For diarrhea syndrome, three symptoms (diarrhea, loose stools, urgent need for defecation) will each be measured on a seven point Likert scale (0=no symptom, 6=most severe symptom). The three values will be averaged to provide one value which will represent diarrhea syndrome.
Indigestion syndrome | 1 year
  The average increase among all subjects using the Gastrointestinal Symptom Rating Scale. For indigestion syndrome, five symptoms (nausea, stomach rumbling, feeling bloated, burping, and passing gas) will each be measured on a seven point Likert scale (0=no symptom, 6=most severe symptom). The five values will be averaged to provide one value which will represent indigestion syndrome.
Acid reflux syndrome | 1 year
  The average increase among all subjects using the Gastrointestinal Symptom Rating Scale. For acid reflux syndrome, two symptoms (heart burn and acid reflux) will each be measured on a seven point Likert scale (0=no symptom, 6=most severe symptom). The two values will be averaged to provide one value which will represent acid reflux syndrome.
Abdominal pain syndrome | 1 year
  The average increase among all subjects using the Gastrointestinal Symptom Rating Scale. For abdominal pain syndrome, two symptoms (stomach ache and hunger pains) will each be measured on a seven point Likert scale (0=no symptom, 6=most severe symptom). The two values will be averaged to provide one value which will represent abdominal pain syndrome.

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey E Friedman, MD, Principal Investigator — University of Florida
Locations (1):
- University of Florida, Gainesville, Florida, United States

IPD SHARING:
Plan to Share IPD: No